CLINICAL TRIAL: NCT06382935
Title: Effects of Minimally Non-surgical Periodontal Treatment Versus Quadrantwise Subgingival Instrumentations on miRNome in Gingival Tissues
Brief Title: Impact of Non-surgical Periodontal Treatment of miRNome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Gaetano Isola, Associate Professor, University of Catania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34-24
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Non-surgical periodontal treatment Subgingival biofilm ultrasonic debridement with MINST or Q-SI
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST non surgical periodontal treatment (Experimental): Periodontitis patients treated by means of MINST. Patients were treated with non-surgical MINST periodontal treatment in a single session.
  Interventions: Other: Probin Pocket Depth reduction
- Q-SI non surgical periodontal treatment (Active Comparator): Periodontitis patients treated by means of Q-SI. Patients were treated with non-surgical quadrantwise periodontal treatment in 4 sessions, 1 session per week.
  Interventions: Other: Probin Pocket Depth reduction

INTERVENTIONS:
Other: Probin Pocket Depth reduction — Probin Pocket Depth reduction in millimetres before and after treatment

SUMMARY:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment by means of minimally invasive approach MINST or Q-SI (quadrantwise) approach in subjects with periodontitis on miRNome in gingival crevicular fluid

DETAILED DESCRIPTION:
A double-blind randomized-controlled clinical trial is conducted in order to evaluate the impact of non-surgical periodontal treatment in subjects with periodontitis.

60 patients: 30 with periodontitis and 30 healthy controls. All the patients are assessed for clinical, periodontal, blood following of minimally invasive approach MINST or Q-SI (quadrantwise).

Measurements are taken before and after initial periodontal treatment in the periodontal subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Periodontitis

Exclusion Criteria:

* Periodontal treatment
* Use of antibiotics, NSAIDs, and immunosuppressants during the last 6 months
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-09-22 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Probing Pocket Depth | 6-months
  Reduction in Probing Pocket Depth after treatnebt

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Catania
Locations (1):
- AOU Policlinico G. Rodolico, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study results
Supporting Information: Study Protocol
Time Frame: 1-year
Access Criteria: Pubmed
URL: https://pubmed.ncbi.nlm.nih.gov/